CLINICAL TRIAL: NCT03741309
Title: Comparison of Clinical Efficacy of a Dentifrice Containing 5% Fluoro Calcium Phosphosilicate to a Dentifrice Containing Calcium Sodium Phosphosilicate and to a Placebo on Dentinal Hypersensitivity : a Randomized Clinical Trial
Brief Title: Comparison of Clinical Efficacy of a Dentifrice Containing 5% Fluoro Calcium Phosphosilicate to a Dentifrice Containing Calcium Sodium Phosphosilicate on Dentinal Hypersensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Collaborators: Group Pharma (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Head and Professor, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/Ph.D/5/2016-2017N
Record Dates: First submitted 2018-11-11; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Dentinal Hypersensitivity
Keywords: dentinal hypersensitivity; visual analog scale

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): dentifrice containing 5% fluorocalcium phospho silicate prescribed and VAS score assessed at Baseline, 2 weeks, 6 weeks.
  Interventions: Other: 5% fluorocalcium phosphosilicate dentifrice
- Group II (Sham Comparator): dentifrice containing Calcium sodium phosphosilicate prescribed and VAS score assessed at Baseline, 2weeks, 6 weeks .
  Interventions: Other: Calcium sodium phosphosilicate
- Group III (Placebo Comparator): dentifrice without the active ingredient prescribed and VAS score assessed at Baseline, 2weeks, 6 weeks.
  Interventions: Other: Placebo dentrifice

INTERVENTIONS:
Other: 5% fluorocalcium phosphosilicate dentifrice — dentifrice containing 5% fluorocalcium phosphosilicate and VAS score assessed at Baseline, 2 weeks, 6 weeks.
  Arms: Group I
Other: Calcium sodium phosphosilicate — Calcium sodium phosphosilicatand VAS score assessed at Baseline, 2weeks, 6 weeks.
  Arms: Group II
Other: Placebo dentrifice — placebo dentifrice and VAS score assessed at Baseline, 2weeks, 6 weeks.
  Arms: Group III

SUMMARY:
Aim of this study was to assess and compare the efficacy of a dentifrice containing 5% fluoro calcium phosphosilicate and dentifrice containing calcium sodium phosphosilicate on Dentinal Hypersensitivity (DH) compared to a placebo over a period of 6 weeks.

DETAILED DESCRIPTION:
A total of 131 subjects were divided into 3 groups randomly. Group I was given the dentifrice containing 5% fluoro calcium phosphosilicate ,Group II was given the dentifrice containing calcium sodium phosphosilicate and group III was given placebo. Sensitivity scores (VAS score) were recorded at baseline, 2 weeks, 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The volunteers selected at baseline were in good general health and should have at least 20 natural permanent teeth and history of hypersensitivity to hot, cold, sour stimuli on at least two teeth with a VAS score of ≥4.

Exclusion Criteria:

* Patients with active cervical caries or deep abrasion requiring cervical filling, chipped teeth or fractured cusps, tender tooth in same quadrant as the hypersensitive teeth, Subjects using any type of desensitizing paste or desensitizing therapy for last 6 months, Pregnant/ lactating women or subjects with history of chronic use of anti-inflammatory and analgesic medications were excluded.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-24 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale score for Dentinal Hypersensitivity | Change in VAS score from Baseline to 6 weeks
  Based on a 10-cm VAS score which was used to measure tooth sensitivity, a pain-free response was allotted a score of zero whereas a score of 10 was given to subjects with excruciating pain or discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Avani R Pradeep, MDS, Principal Investigator — GDCRI, Bangalore, INDIA
Locations (1):
- Department of Periodontics, GDCRI Bangalore, Bangalore, Karnataka, India